CLINICAL TRIAL: NCT04120402
Title: A Phase 2, Randomized, Double-Blind, Vehicle-Controlled Study Evaluating the Safety, Efficacy and Pharmacokinetics of Single Dose EP-104IAR for 24 Weeks in Patients With Osteoarthritis of the Knee
Brief Title: Study to Evaluate the Efficacy and Safety of EP-104IAR in Patients With Osteoarthritis of the Knee
Acronym: SPRINGBOARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eupraxia Pharmaceuticals Inc. (Industry)
Collaborators: NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP-104IAR-201
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to received either EP-104IAR or placebo (vehicle) in a parallel group fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EP-104IAR 25 mg (Experimental): A single use intra-articular injection containing 25 mg of EP-104IAR
  Interventions: Drug: EP-104IAR 25 mg
- Placebo (vehicle) (Placebo Comparator): A single use intra-articular injection containing no active ingredients
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: EP-104IAR 25 mg — Single 5 mL intra-articular injection
  Arms: EP-104IAR 25 mg
Drug: Vehicle — Single 5 mL intra-articular injection
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and pharmacokinetics (PK) of EP-104IAR in patients with osteoarthritis (OA) of the knee

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single injection, 24-week study to evaluate the safety, efficacy and PK of EP-104IAR in subjects with osteoarthritis knee pain

Following screening and baseline assessments to determine eligibility, each participant will receive a single IA injection of either EP-104IAR or placebo (vehicle). Participants will be followed up for 24 weeks following the injection for safety, PK and efficacy assessments.

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females, aged ≥40 years
* Body Mass Index (BMI) ≤ 40.0 kg/m2
* Diagnosis of primary OA of the Index knee, with symptoms present for at least 6 months
* OA severity Grade 2 or 3 (based on Kellgren Lawrence Grading Scale)
* Unsatisfactory pain relief from at least 2 prior standard OA treatments
* Qualifying pain in the Index knee during the baseline period
* Ambulatory (without the need for a cane/other walking aide)
* Female subjects willing to use highly effective birth control methods to prevent pregnancy
* Willing and able to comply with study procedures and restrictions, including abstaining from use of restricted medications.

Key Exclusion Criteria:

* OA of the Index knee due to acute injury or trauma, or unstable joint
* X-ray evidence of chondrocalcinosis
* Diagnosed or suspected ipsilateral hip OA
* Knee pain that is not attributable to OA of the knee
* Any other disorders that impact mobility, strength or sensation, or are a co-existent source of pain or inflammation that interfere with assessment of knee pain and function
* History of infection in the Index knee
* Skin breakdown on the Index knee where the injection will take place
* Total Knee Replacement, or any other surgery (including arthroscopy) for the Index knee within prior 12 months, or planned surgery during the study
* Total Knee Replacement Surgery of the non-Index knee within prior 6 months, or planned surgery (any location) during the study that would require a restricted medication
* IA injection of corticosteroids in any joint within prior 3 months or IA injection of extended-release corticosteroids in any joint within prior 6 months
* IA injection in the Index knee of platelet rich plasma, or other prolotherapy within prior 3 months, or hyaluronic acid within prior 6 months
* Recent, current or planned use of corticosteroids for any indication (except for permitted uses)
* Recent, current or planned use of prohibited medications (including analgesics, marijuana, investigational drugs and devices, immunosuppressive therapy), or unwilling or unable to stop using prohibited medications during the study.
* Conditions including: sarcoidosis, amyloidosis, osteomyelitis, Cushing's Syndrome, hepatic or renal disease, Psychotic disorder, bipolar disorder, symptomatic depressive or anxiety disorders.
* Current malignancy of any type, or history of a malignancy within prior 12 months
* Active or quiescent systemic fungal, bacterial (including tuberculosis) viral (including HIV, Hepatitis B or C) or parasitic infections, or ocular herpes simplex, or any recent infection requiring IV or oral antibiotics
* Laboratory results indicative of adrenal insufficiency, diabetes or renal or hepatic disease.
* Positive urine drug screen for a substance of abuse
* Females who are pregnant, lactating
* Known or suspected hypersensitivity or contraindication to ingredients in the study drug

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Malone, Study Director — Eupraxia Pharmaceuticals
Locations (12):
- Czechia (3):
  - CCR Brno, s.r.o, Brno
  - CCR Czech a.s, Pardubice
  - CCR Prague, s.r.o, Prague
- Denmark (4):
  - The Parker Institute, Frederiksberg Hospital, Frederiksberg
  - Sanos Clinic Nordjylland, Gandrup
  - Sanos Clinic Herlev, Herlev
  - Sanos Clinic Syddanmark, Vejle
- Poland (5):
  - NZOZ BIF-MED s.c, Bytom
  - Somed CR, Lodz
  - Medyczne Centrum Hetmańska, Poznan
  - DC-MED, Swidnica
  - Somed CR, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malone A, Kowalski MM, Helliwell J, Lynggaard Boll S, Rovsing H, Moriat K, Castillo Mondragon A, Li Y, Prener Miller C, Reinstrup Bihlet A, Dobek C, Peck V, Wilmink M, Simon LS, Conaghan PG. Efficacy and safety of a diffusion-based extended-release fluticasone propionate intra-articular injection (EP-104IAR) in knee osteoarthritis (SPRINGBOARD): a 24-week, multicentre, randomised, double-blind, vehicle-controlled, phase 2 trial. Lancet Rheumatol. 2024 Dec;6(12):e860-e870. doi: 10.1016/S2665-9913(24)00223-6. Epub 2024 Oct 11. PMID 39401503

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EP-104IAR 25 mg | Placebo (Vehicle)
Started | 163 | 155
Completed | 156 | 148
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population consisted of all subjects who were both randomized to and received treatment. Analysis was conducted allocating subjects to the treatment to which they were randomized, irrespective of what was actually received. The safety population consisted of all randomized subjects who were administered a dose of study drug. The subjects in this group were analyzed based on the treatment they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | EP-104IAR 25 mg | Placebo (Vehicle) | Total
Number analyzed (Participants) | 163 | 155 | 318
Age, Categorical [Count of Participants; unit: Participants] — Population: The analysis population is the intent to treat population of 318 patients in total. Out of the 318 patients 163 patients were in the EP-104IAR 25mg arm and 155 patients were in the Placebo (Vehicle) arm.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 91 | 89 | 180
    >=65 years | 72 | 66 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.31) | 63.2 (9.37) | 63.6 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 89 | 183
  Male | 69 | 66 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 161 | 152 | 313
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 162 | 153 | 315
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czechia | 40 | 35 | 75
  Denmark | 85 | 84 | 169
  Poland | 38 | 36 | 74

OUTCOME MEASURES:

1. Primary Outcome: Difference in Change From Baseline Between EP-104IAR and Vehicle in WOMAC Pain Subscale
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale (scores scaled 0-10, with 10 being the worst). Least squares mean from a mixed model for repeated measures (MMRM) for change from baseline with fixed effects for site, treatment, week, treatment-by-week interaction; random effect for subject; and covariate baseline WOMAC pain score.
Time Frame: 12 weeks
Population: The intention-to-treat (ITT) population consists of all subjects who were both randomized to and received treatment. Analysis was conducted allocating subjects to the treatment to which they were randomized, irrespective of what was actually received.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | EP-104IAR 25 mg | Placebo (Vehicle)
Number analyzed (Participants) | 163 | 155
score on a scale | -2.89 (0.166) | -2.23 (0.171)
Statistical Analysis 1: Comparison: EP-104IAR 25 mg vs Placebo (Vehicle); Test type: Superiority; p = 0.004, ANCOVA

2. Secondary Outcome: Difference in Change From Baseline Between EP-104IAR and Vehicle in WOMAC Function Subscale
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale (scores scaled 0-10, with 10 being the worst). Function subscale includes questions related to the physical functioning of osteoarthritis e.g. stair use, standing, walking etc. From a mixed model for repeated measures (MMRM) for change from baseline with fixed effects for site, treatment, week, treatment-by-week interaction; random effect for subject; and covariate baseline WOMAC function score.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | EP-104IAR 25 mg | Placebo (Vehicle)
Number analyzed (Participants) | 163 | 155
score on a scale | -2.59 (0.161) | -2.04 (0.166)
Statistical Analysis 1: Comparison: EP-104IAR 25 mg vs Placebo (Vehicle); Test type: Superiority; p = 0.014, ANCOVA

3. Secondary Outcome: Difference Between EP-104IAR and Vehicle in the Area Under the Curve (AUC) of WOMAC Pain Subscale
Description: Area under the curve in change from baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale (scores scaled 0-10, with 10 being the worst) from Week 0 to Week 12 was calculated on a per-individual basis using the linear trapezoidal rule. AUC was normalized to account for subjects whose actual days and nominal days at Week 12 differed. Treatments were compared using an ANCOVA model containing site; individual baseline WOMAC Pain; and treatment group as covariates.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale multiplied by days
Arm/Group | EP-104IAR 25 mg | Placebo (Vehicle)
Number analyzed (Participants) | 163 | 155
score on a scale multiplied by days | -235.67 (11.769) | -166.78 (12.169)
Statistical Analysis 1: Comparison: EP-104IAR 25 mg vs Placebo (Vehicle); Test type: Superiority; p < 0.001, ANCOVA

4. Secondary Outcome: Difference in Change From Baseline Between EP-104IAR and Vehicle in WOMAC Pain Subscale
Description: as for outcome 1
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | EP-104IAR 25 mg | Placebo (Vehicle)
Number analyzed (Participants) | 163 | 155
score on a scale | -2.26 (0.171) | -2.11 (0.175)
Statistical Analysis 1: Comparison: EP-104IAR 25 mg vs Placebo (Vehicle); Test type: Superiority; p = 0.518, ANCOVA

5. Secondary Outcome: Difference Between EP-104IAR and Vehicle in OMERACT-OARSI Strict Responders
Description: Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) strict responders are defined as at least 50% improvement (decrease from baseline) in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain or function subscales (scores scaled 0-10, with 10 being the worst) and an absolute change of at least 2 in the respective score. Patients who discontinued prior to Week 12 were considered non-responders.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EP-104IAR 25 mg | Placebo (Vehicle)
Number analyzed (Participants) | 163 | 155
Participants | 87 | 61
Statistical Analysis 1: Comparison: EP-104IAR 25 mg vs Placebo (Vehicle); Test type: Superiority; p = 0.028, Fisher Exact

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were summarized and analyzed for safety evaluations i.e, events which occurred from the time of the EP-104IAR or vehicle injection procedure until the Week 24/End-of-Study/Early Exit Visit.
Arm/Group | EP-104IAR 25 mg | Placebo (Vehicle)
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/155
Serious Adverse Events (participants affected / at risk) | 4/163 | 1/155
Other Adverse Events (participants affected / at risk) | 76/163 | 68/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EP-104IAR 25 mg (N=163) | Placebo (Vehicle) (N=155)
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EP-104IAR 25 mg (N=163) | Placebo (Vehicle) (N=155)
Nasopharyngitis (Infections and infestations) | 14 (16) | 12 (15)
COVID-19 (Infections and infestations) | 14 (14) | 14 (14)
Influenza (Infections and infestations) | 6 (6) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 (38) | 23 (26)
Influenza like illness (General disorders) | 4 (5) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may not present or publish partial or complete study results individually without the Sponsor's agreement.

Any manuscript or abstract proposed by the Investigators must be reviewed and approved in writing by the Sponsor before submission for publication. Names of all Investigators participating in the study will be included in the publication.

DOCUMENTS (2):
  • Study Protocol (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT04120402/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT04120402/SAP_001.pdf